CLINICAL TRIAL: NCT06035809
Title: The Effects of Sensory Motor Arousal Regulation Treatment (SMART) on Adults With PTSD
Brief Title: Sensory Motor Arousal Regulation Treatment (SMART) Study
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ruth Lanius, MD, PhD, Professor of Psychiatry, Harris-Woodman Chair, University of Western Ontario, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ReDA: 12919; 121855 (Other: Western Research Ethics Board)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: PTSD; Post-traumatic Stress Disorder
Keywords: PTSD; Post-traumatic Stress Disorder; Body-based trauma therapy; Movement-based trauma therapy; Sensory-motor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a study investigating SMART as an intervention for symptoms of PTSD. Participants will be randomized to one of two conditions: SMART or Wait List (i.e., delayed treatment), and both groups will be assessed at 3 time points.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to which treatment arm a participant was assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active SMART (Experimental): Participants in the active SMART condition will complete 8 individual, 1-hour, weekly sessions of SMART with a therapist, as well as pre-treatment, post-treatment and 3-month follow-up assessments.
  Interventions: Behavioral: SMART
- Wait List (No Intervention): Participants in the Wait List condition will receive no treatment for approximately 8 weeks, and they will be asked to complete pre-wait list, post-wait list and 3-month follow-up assessments. After all assessments have been completed, this group will be offered the same 8 individual, 1-hour, weekly sessions of SMART (no further assessments needed).

INTERVENTIONS:
Behavioral: SMART — A movement and body-based intervention in which participants are encouraged to explore the use of sensory equipment, which may help reduce symptoms related to psychological trauma/PTSD. Sensory equipment includes exercise balls, mini-trampoline, weighted blankets, and a hammock swing.
  Arms: Active SMART

SUMMARY:
This study will investigate whether a movement and body-based treatment can benefit adults with Post-traumatic Stress Disorder (PTSD). The treatment is called Sensory Motor Arousal Regulation Treatment, or "SMART", and study participation involves 8 sessions of SMART, as well as pre-treatment, post-treatment, and 3-month follow-up assessments.

DETAILED DESCRIPTION:
This study will investigate the use of SMART (Sensory Motor Arousal Regulation Treatment) with adults experiencing symptoms related to PTSD (Post-Traumatic Stress Disorder). In addition to the more well-known symptoms of PTSD (e.g., intrusive memories, avoidance, hypervigilance, and emotion dysregulation), chronic traumatic stress seems to overwhelm the brain's capacity to make sense of sensory information, affecting how traumatized people experience their own bodies and their surroundings. SMART builds on the sensory integration theory of intentionally engaging the senses via movement, touch, body awareness, and balance. The SMART protocol has been used effectively to treat children who have experienced psychological trauma, and the investigators will be investigating its use with adults. Participants enrolled in the study will be randomly assigned to one of two treatment conditions - i) SMART, or ii) wait list (i.e., delayed treatment). Study participation will involve 8, 1-hour sessions of SMART, as well as pre-treatment, post-treatment, and 3-month follow-up assessments. For those assigned to the wait list condition, the same 8 SMART sessions will be offered after the 3-month follow-up assessment is complete, with no further assessment required.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18-65
2. A primary diagnosis of PTSD as determined by our pre-treatment assessment
3. Ability to provide informed consent
4. Fluency in written and spoken English (to be able to complete assessments)

Exclusion Criteria:

1. any implants, conditions, etc. that do not comply with 7T (Tesla) fMRI research safety standards (e.g., pacemaker, pregnancy/possible pregnancy)
2. history of significant head injury/lengthy loss of consciousness (e.g., a Glasgow Coma Scale Score < 15 at the time of incident as assessed retrospectively by participant)
3. significant untreated medical illness
4. history of neurological or neurodevelopmental disorder
5. history of any pervasive developmental disorder
6. lifetime bipolar or psychotic disorder
7. alcohol/substance abuse or dependence within the last 3 months
8. extensive narcotic use (e.g., fentanyl, oxycodone, etc.)
9. anyone who would not be suitable for short-term treatment (as determined by our pre-treatment assessment)
10. suicide attempt in last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS) score from pre-treatment to post-treatment assessment. | 8 weeks
  Gold standard, clinician-administered PTSD assessment tool; min. score=0, max.=80, with higher scores representing greater PTSD symptoms
Change in Clinician Administered PTSD Scale (CAPS) score from post-treatment to 3-month follow-up assessment. | 12 weeks
  Gold standard, clinician-administered PTSD assessment tool; min. score=0, max.=80, with higher scores representing greater PTSD symptoms

SECONDARY OUTCOMES:
Change in Multidimensional Assessment of Interoceptive Awareness (MAIA-II) score from pre-treatment to post-treatment assessment. | 8 weeks
  A state-trait, self-report questionnaire with 32 items to measure multiple dimensions of interoception (e.g., awareness of the senses). Higher scores indicate beneficial self-reported interoception.
Change in Multidimensional Assessment of Interoceptive Awareness (MAIA-II) score from post-treatment to 3-month follow-up assessment. | 12 weeks
  A state-trait, self-report questionnaire with 32 items to measure multiple dimensions of interoception (e.g., awareness of the senses). Higher scores indicate beneficial self-reported interoception.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lanius, MD, PhD, Principal Investigator — Lawson Health Research/Western University/LHSC
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only coded data will be shared with co-investigators who are registered with the study's ethics board application.

REFERENCES:
- [Background] Finn H, Warner E, Price M, Spinazzola J. The Boy Who Was Hit in the Face: Somatic Regulation and Processing of Preverbal Complex Trauma. J Child Adolesc Trauma. 2017 Jun 29;11(3):277-288. doi: 10.1007/s40653-017-0165-9. eCollection 2018 Sep. PMID 32318157
- [Background] Lanius RA, Frewen PA, Tursich M, Jetly R, McKinnon MC. Restoring large-scale brain networks in PTSD and related disorders: a proposal for neuroscientifically-informed treatment interventions. Eur J Psychotraumatol. 2015 Mar 31;6:27313. doi: 10.3402/ejpt.v6.27313. eCollection 2015. PMID 25854674
- [Background] Harricharan S, Nicholson AA, Densmore M, Theberge J, McKinnon MC, Neufeld RWJ, Lanius RA. Sensory overload and imbalance: Resting-state vestibular connectivity in PTSD and its dissociative subtype. Neuropsychologia. 2017 Nov;106:169-178. doi: 10.1016/j.neuropsychologia.2017.09.010. Epub 2017 Sep 11. PMID 28911803
- [Background] Lanius RA, Terpou BA, McKinnon MC. The sense of self in the aftermath of trauma: lessons from the default mode network in posttraumatic stress disorder. Eur J Psychotraumatol. 2020 Oct 23;11(1):1807703. doi: 10.1080/20008198.2020.1807703. PMID 33178406
- [Background] Warner, E., Westcott, A., Cook, A., & Finn, H. (2020). Transforming trauma in children and adolescents: An embodied approach to somatic regulation, trauma processing, and attachment-building. North Atlantic Books.